CLINICAL TRIAL: NCT01686386
Title: A Phase I/II Study of Bendamustine, Lenalidomide and Low-dose Dexamethasone, (BdL) for the Treatment of Patients With Relapsed Myeloma.
Brief Title: Study of Bendamustine, Lenalidomide and Low-dose Dexamethasone, for the Treatment of Patients With Relapsed Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-GIMEMA/GISL430; 2010-018336-40 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-09-18 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Multiple Myeloma; Lenalidomide; Bendamustine
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bendamustine Hydrochloride; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation benda lena dexa (Experimental): Phase I: Participants will be treated in groups (cohorts) of three to six subjects per cohort, according to a modified Fibonacci design. The dose of Bendamustine and Lenalidomide (from 0 to 5) will be increased from one cohort to the next. Regardless of the treatment cohort, participants will receive treatment in cycles lasting 28 days. In the first phase of the study, the dose of B and L given with will be gradually escalated to reach the MTD.
  Phase II: Dexamethasone will be given in combination with the MTD of Bendamustine and Lenalidomide in cycles lasting 28 days.
  Interventions: Drug: Bendamustine; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Phase I: dose escalation of Bendamustine Phase II: Dexamethasone will be given in combination with the MTD of Bendamustine and Lenalidomide in cycles lasting 28 days.
Drug: Lenalidomide — Phase I: dose escalation of Lenalidomide Phase II: Dexamethasone will be given in combination with the Maximum Tolerated Dose (MTD) of Bendamustine and Lenalidomide in cycles lasting 28 days.
Drug: Dexamethasone — Phase I and Phase II Dexamethasone fixed dose 40 mg/die

SUMMARY:
This is an open Label, Phase I/II, multicenter study. In the first phase it defines the maximum tolerated dose (MTD) of Bendamustine (B) given in combination with Lenalidomide (L) and low-dose Dexamethasone (d) and in the second phase it evaluates the antitumour activity of Bendamustine, Lenalidomide and Low-dose Dexamethasone (BdL) given in combination, in relapsed multiple myeloma patients.

DETAILED DESCRIPTION:
Multiple myeloma is a B-cell malignancy resulting from the monoclonal proliferation of plasma cells within the bone marrow. According to the American Cancer Society, 14,600 new cases of multiple myeloma will be diagnosed in 2002, and these will account for approximately 1% of all new cancer cases. Multiple myeloma will contribute to 2% of all cancer deaths this year; an estimated 10,800 deaths will occur overall. The disease is more prevalent in men and is twice as common in African-Americans as in Caucasians. Multiple myeloma is commonly thought of as a disease of older patients; the median age at diagnosis is 68 years, and the incidence increases more than 4%/year in those older than 85 years. The median survival with standard treatment is only 3 years.

Therapeutic options for patients with multiple myeloma (MM) are rapidly changing. The emergence of two highly active novel agents, bortezomib and lenalidomide, have dramatically changed the landscape of treatment options and have improved outcomes for many patients. Combinations of conventional agents with novel agents have also demonstrated significant efficacy for patients with newly diagnosed and relapsed myeloma. Among the conventional agents that are being explored is the bifunctional alkylator agent bendamustine, which has demonstrated single-agent activity and activity with novel agents.

Lenalidomide is a new immunomodulating agent effective in multiple myeloma, especially when associated with dexamethasone or melphalan and prednisone. The role of lenalidomide in the treatment of relapsed/refractory patients with MM has been established and current research is focused on the combination of lenalidomide with chemotherapy to further improve results.

Bendamustine is a bi-functional alkylating agent with a purine- like benzimidazole ring that has been administered successfully to patients with MM. In vitro studies showed that bendamustine possesses a unique profile of activity, which was clearly divergent from other common nitrogen mustard drugs. Bendamustine and prednisone in newly diagnosed MM patients results in superior complete response rate, prolonged time to treatment failure and improved quality of life compared to treatment with melphalan and prednisone. The role of bendamustine, thalidomide and prednisolone (BPT) in patients with relapsed or refractory diseases stage II/III has been investigated by the East German Study group of Hematology and Oncology (OSHO). The response rate was higher than 80%.

Despite the impressive efficacy of the lenalidomide/dexamethasone in relapsed MM, treated patients will eventually relapse (median Time to Progression (TTP) is expected to be nearly a year according the results of the two phase III randomized studies). Combination with an effective novel agent as bendamustine could further increase both the response rate and the TTP of lenalidomide/dexamethasone and induce durable responses in relapsed or refractory MM patients. The identification of an appropriate lenalidomide dose to be adopted in combination with bendamustine and dexamethasone and the generation of exploratory data on the efficacy of this novel combination appears to be important in terms of future development of even more effective treatments of MM.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Men and women age ≥ 18 years
* Female subjects are either post-menopausal or surgically sterilized or willing to use 2 simultaneous methods of contraception
* Male patients must agree to use a latex condom during sexual contact with females of childbearing potential throughout the study and for at least 28 days following discontinuation of lenalidomide;
* Confirmed diagnosis of Multiple Myeloma with measurable disease .Patients with evidence of relapsed disease after more than 1 and equal but not more than 3 prior lines of therapy.
* ECOG Performance Status 0 - 2
* Required baseline haematology and chemistry parameters

Exclusion Criteria:

* Myocardial infarction within 6 months prior to enrollment or has NYHA class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Female subjects either pregnant or breast-feeding (negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result)
* Patients have received other investigational drugs with 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Any of the following laboratory abnormalities:

Absolute neutrophil count (ANC) <1,000 /μl (1x109 /L) Untransfused platelet count < 50,0000cell/μl (50x109 /L) Serum SGOT/AST or SGPT/ALT > 2.0 upper limit of normal (ULN) Total bilirubin > 2.0 mg/dL Renal insufficiently (serum creatinine level > 2.5 mg/dl or Creatinine clearance < 30 mL/min calculated by Cockcroft-Gault estimation)

* Patients with active infections are ineligible.
* Patients who are HIV positive are ineligible.
* Patients with active leptomeningeal involvement are ineligible.
* Patients with a history of previous CSF tumor involvement without symptoms or signs are eligible provided the CSF is now free of disease on lumbar puncture, and MRI of the brain shows no tumor involvement.
* History of other malignancies within 3 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or breast, low grade, early stage localized prostate cancer treated surgically with curative intent (TNM stage of T1a or T1b),
* Patients with uncontrolled insulin-dependent diabetes mellitus or uncompensated major thyroid or adrenal dysfunction are ineligible.
* Patients with an ECOG performance status of > 2 are ineligible.
* Malabsorption syndrome or uncontrolled gastrointestinal toxicities
* Clinically significant pleural effusion in the previous 12 months or current ascitis
* Clinically-significant coagulation or platelet function disorder
* Intolerance to bendamustine and/or lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Phase I:Determination of Maximum Tolerated Dose | up to 28 days during first cycle
  In the first phase of the study, the dose of Bendamustine and Lenalidomide given with will be gradually escalated to reach the Maximum Tolerated Dose. The Maximum Tolerated Dose of Bendamustine and Lenalidomide will be evaluated during the first course (cycle 1) of Bendamustine Dexamethasone Lenalidomide (BdL) administered
Phase I:Determination of occurrence rate of AE/SAEs | up to 28 day (during the first cycle 1of BdL administered)
  To assess the Safety and Toxicity of the Bendamustine,Dexamethasone and Lenalidomide (BdL) regimen
Phase II: Overall Response Rate (ORR) | An avarage of 6 months (after 6 cycles of therapy)
  To assess the antitumour activity of the BdL regimen, in term of Complete response, Partial response and Stable disease, according to the best schedule identified during Phase I.

SECONDARY OUTCOMES:
Phase I: Assessment of the preliminary antineoplastic properties of the BdL | after an avarage of 6 months
  To explore the preliminary antitumor activity of drug combination in patients with relapsed MM
Phase II: AE/SAEs | Every 28 days (during all cycles)
  To define the safety profile of the treatment assessing the occurrence rate and the severity
Phase II:Determination of the response rates | Assessed after 6 months
  To assess Partial Response and Complete Response rates
Phase II:Time to Event parameters | avarage 6 months
  To evaluate the efficacy of the BdL regimen in patients with relapsed MM, in terms of Progression-Free Survival, Time to Progression, Time to Response, Duration of Response ,Overall Survival(PFS, TTP, TTR, DR, OS)

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Morabito, MD, Study Chair — Unità Operativa Complessa di Ematologia- Stabilimento Ospedaliero Annunziata - Azienda Ospedaliera di Cosenza
Locations (1):
- U. O. C. Ematologia - Azienda Ospedaliera Cosenza, Cosenza, Cosenza, Italy

REFERENCES:
- [Background] Munshi NC, Tricot G, Barlogie B. Plasma cell neoplasms. In: DeVita VT Jr, Hellman S, Rosenberg SA, eds. Cancer: principles and practice of oncology, 6th ed. Philadelphia, PA: Lippincott Williams & Wilkins, 2001:2465-99.
- [Background] Jemal A, Thomas A, Murray T, Thun M. Cancer statistics, 2002. CA Cancer J Clin. 2002 Jan-Feb;52(1):23-47. doi: 10.3322/canjclin.52.1.23. PMID 11814064
- [Background] Durie BG. The epidemiology of multiple myeloma. Semin Hematol. 2001 Apr;38(2 Suppl 3):1-5. doi: 10.1016/s0037-1963(01)90087-3. PMID 11309701
- [Background] Kishi Y, Oki Y, Machida U. Thalidomide in multiple myeloma. N Engl J Med. 2000 Mar 30;342(13):975; author reply 975-6. doi: 10.1056/NEJM200003303421313. No abstract available. PMID 10744492
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Palumbo A, Falco P, Corradini P, Falcone A, Di Raimondo F, Giuliani N, Crippa C, Ciccone G, Omede P, Ambrosini MT, Gay F, Bringhen S, Musto P, Foa R, Knight R, Zeldis JB, Boccadoro M, Petrucci MT; GIMEMA--Italian Multiple Myeloma Network. Melphalan, prednisone, and lenalidomide treatment for newly diagnosed myeloma: a report from the GIMEMA--Italian Multiple Myeloma Network. J Clin Oncol. 2007 Oct 1;25(28):4459-65. doi: 10.1200/JCO.2007.12.3463. Epub 2007 Sep 4. PMID 17785703
- [Background] Anger G, Hesse P, Baufeld H. [Treatment of multiple myeloma with a new cytostatic agent: gamma-l-methyl-5-bis-(beta-chlorethyl)-amino-benzimidazolyl-(2)-butyric acid hydrochloride]. Dtsch Med Wochenschr. 1969 Nov 28;94(48):2495-500. doi: 10.1055/s-0028-1110470. No abstract available. German. PMID 4903552
- [Background] Leoni LM, Bailey B, Reifert J, Bendall HH, Zeller RW, Corbeil J, Elliott G, Niemeyer CC. Bendamustine (Treanda) displays a distinct pattern of cytotoxicity and unique mechanistic features compared with other alkylating agents. Clin Cancer Res. 2008 Jan 1;14(1):309-17. doi: 10.1158/1078-0432.CCR-07-1061. PMID 18172283
- [Background] Ponisch W, Mitrou PS, Merkle K, Herold M, Assmann M, Wilhelm G, Dachselt K, Richter P, Schirmer V, Schulze A, Subert R, Harksel B, Grobe N, Stelzer E, Schulze M, Bittrich A, Freund M, Pasold R, Friedrich T, Helbig W, Niederwieser D; East German Study Group of Hematology and Oncology (OSHO). Treatment of bendamustine and prednisone in patients with newly diagnosed multiple myeloma results in superior complete response rate, prolonged time to treatment failure and improved quality of life compared to treatment with melphalan and prednisone--a randomized phase III study of the East German Study Group of Hematology and Oncology (OSHO). J Cancer Res Clin Oncol. 2006 Apr;132(4):205-12. doi: 10.1007/s00432-005-0074-4. Epub 2006 Jan 10. PMID 16402269
- [Background] Ponisch W, Rozanski M, Goldschmidt H, Hoffmann FA, Boldt T, Schwarzer A, Ritter U, Rohrberg R, Schwalbe E, Uhlig J, Zehrfeld T, Schirmer V, Haas A, Kreibich U, Niederwieser D; East German Study Group of Haematology and Oncology (OSHO). Combined bendamustine, prednisolone and thalidomide for refractory or relapsed multiple myeloma after autologous stem-cell transplantation or conventional chemotherapy: results of a Phase I clinical trial. Br J Haematol. 2008 Oct;143(2):191-200. doi: 10.1111/j.1365-2141.2008.07076.x. Epub 2008 Aug 24. PMID 18752593
- [Background] List A, Kurtin S, Roe DJ, Buresh A, Mahadevan D, Fuchs D, Rimsza L, Heaton R, Knight R, Zeldis JB. Efficacy of lenalidomide in myelodysplastic syndromes. N Engl J Med. 2005 Feb 10;352(6):549-57. doi: 10.1056/NEJMoa041668. PMID 15703420
- [Background] List A, Dewald G, Bennett J, Giagounidis A, Raza A, Feldman E, Powell B, Greenberg P, Thomas D, Stone R, Reeder C, Wride K, Patin J, Schmidt M, Zeldis J, Knight R; Myelodysplastic Syndrome-003 Study Investigators. Lenalidomide in the myelodysplastic syndrome with chromosome 5q deletion. N Engl J Med. 2006 Oct 5;355(14):1456-65. doi: 10.1056/NEJMoa061292. PMID 17021321
- [Background] Raza A, Reeves JA, Feldman EJ, Dewald GW, Bennett JM, Deeg HJ, Dreisbach L, Schiffer CA, Stone RM, Greenberg PL, Curtin PT, Klimek VM, Shammo JM, Thomas D, Knight RD, Schmidt M, Wride K, Zeldis JB, List AF. Phase 2 study of lenalidomide in transfusion-dependent, low-risk, and intermediate-1 risk myelodysplastic syndromes with karyotypes other than deletion 5q. Blood. 2008 Jan 1;111(1):86-93. doi: 10.1182/blood-2007-01-068833. Epub 2007 Sep 24. PMID 17893227
- [Background] Rajkumar SV, Jacobus S, Callander N et al. Phase III trial of lenalidomide plus high- dose dexamethasone versus lenalidomide plus low-dose dexamethasone in newly diagnosed multiple myeloma (E4A03): A trial coordinated by the Eastern Cooperative Oncology GroupJournal of Clinical Oncology, 2007 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 25, No 18S (June 20 Supplement), 2007.
- [Background] Rajkumar SV, Jacobus S, Callander N et al. A Randomized Trial of Lenalidomide Plus High-Dose Dexamethasone (RD) Versus Lenalidomide Plus Low-Dose Dexamethasone (Rd) in Newly Diagnosed Multiple Myeloma (E4A03): A Trial Coordinated by the Eastern Cooperative Oncology Group.
- [Background] Chanan-Khan A, Miller KC, Musial L, Lawrence D, Padmanabhan S, Takeshita K, Porter CW, Goodrich DW, Bernstein ZP, Wallace P, Spaner D, Mohr A, Byrne C, Hernandez-Ilizaliturri F, Chrystal C, Starostik P, Czuczman MS. Clinical efficacy of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia: results of a phase II study. J Clin Oncol. 2006 Dec 1;24(34):5343-9. doi: 10.1200/JCO.2005.05.0401. Epub 2006 Nov 6. PMID 17088571
- [Background] Cheson BD, Bennett JM, Grever M, Kay N, Keating MJ, O'Brien S, Rai KR. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood. 1996 Jun 15;87(12):4990-7. No abstract available. PMID 8652811
- [Background] Knauf WU, Lissichkov T, Aldaoud A, Liberati A, Loscertales J, Herbrecht R, Juliusson G, Postner G, Gercheva L, Goranov S, Becker M, Fricke HJ, Huguet F, Del Giudice I, Klein P, Tremmel L, Merkle K, Montillo M. Phase III randomized study of bendamustine compared with chlorambucil in previously untreated patients with chronic lymphocytic leukemia. J Clin Oncol. 2009 Sep 10;27(26):4378-84. doi: 10.1200/JCO.2008.20.8389. Epub 2009 Aug 3. PMID 19652068
- [Background] Friedberg JW, Cohen P, Chen L, Robinson KS, Forero-Torres A, La Casce AS, Fayad LE, Bessudo A, Camacho ES, Williams ME, van der Jagt RH, Oliver JW, Cheson BD. Bendamustine in patients with rituximab-refractory indolent and transformed non-Hodgkin's lymphoma: results from a phase II multicenter, single-agent study. J Clin Oncol. 2008 Jan 10;26(2):204-10. doi: 10.1200/JCO.2007.12.5070. Erratum In: J Clin Oncol. 2008 Apr 10;26(11) 1911. PMID 18182663
- [Background] Rummel MJ, von Gruenhagen U, Niederle N, et al: Bendamustine plus rituximab versus CHOP plus rituximab in the first-line treatment of patients with indolent and mantle-cell lymphomas: The first interim results of a randomized phase III study ofthe StiL (Study Group Indolent Lymphomas, Germany). Blood 110:120a, 2007 (abstr 385).
- [Background] Fenk R, Michael M, Zohren F, Graef T, Czibere A, Bruns I, Neumann F, Fenk B, Haas R, Kobbe G. Escalation therapy with bortezomib, dexamethasone and bendamustine for patients with relapsed or refractory multiple myeloma. Leuk Lymphoma. 2007 Dec;48(12):2345-51. doi: 10.1080/10428190701694194. PMID 18067009
- [Background] Palumbo A, Rajkumar SV, Dimopoulos MA, Richardson PG, San Miguel J, Barlogie B, Harousseau J, Zonder JA, Cavo M, Zangari M, Attal M, Belch A, Knop S, Joshua D, Sezer O, Ludwig H, Vesole D, Blade J, Kyle R, Westin J, Weber D, Bringhen S, Niesvizky R, Waage A, von Lilienfeld-Toal M, Lonial S, Morgan GJ, Orlowski RZ, Shimizu K, Anderson KC, Boccadoro M, Durie BG, Sonneveld P, Hussein MA; International Myeloma Working Group. Prevention of thalidomide- and lenalidomide-associated thrombosis in myeloma. Leukemia. 2008 Feb;22(2):414-23. doi: 10.1038/sj.leu.2405062. Epub 2007 Dec 20. PMID 18094721
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Derived] Pozzi S, Gentile M, Sacchi S, Marcheselli R, Corso A, Cocito F, Musto P, Guarini A, Minoia C, Vincelli I, Ria R, Rivolti E, Mele G, Bari A, Mazzone C, Badiali S, Marcheselli L, Palumbo A, Morabito F. Bendamustine, Low-dose dexamethasone, and lenalidomide (BdL) for the treatment of patients with relapsed/refractory multiple myeloma confirms very promising results in a phase I/II study. Leuk Lymphoma. 2017 Mar;58(3):552-559. doi: 10.1080/10428194.2016.1205741. Epub 2016 Jul 21. PMID 27442600